CLINICAL TRIAL: NCT07019597
Title: Non-invasive NESA Neuromodulation Versus Transcutaneous Posterior Tibial Nerve Stimulation for the Treatment of Overactive Bladder
Brief Title: NESA Neuromodulation Versus Transcutaneous Posterior Tibial Stimulation
Acronym: NesaTibial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel David Álamo Arce (Other)
Responsible Party: Sponsor-Investigator, Daniel David Álamo Arce, Proffesor, University of Las Palmas de Gran Canaria
Organization: University of Las Palmas de Gran Canaria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NesaTibial
Record Dates: First submitted 2025-06-02; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Bladder Dysfunction
Keywords: overactive bladder; Transcutaneous neuromodulation; Nesa Non-Invasive Neuromodulation; Posterior tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: A single-blind, randomised controlled trial was conducted.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: Non-invasive neuromodulation NESA (NNG group) (Experimental): Group 1: Non-invasive NESA® Neuromodulation (NNG) using NESA (Applied superficial stimulation, acronym in spanish) device with same-day exercise and education by providing common, non-individualised written instructions, such as dietary and social advice.
  NNG was performed with the patient supine, using NESA technology with gloves and anklets, with a total of 24 electrodes plus a directional electrode for global neuromodulation; NESA is a non-invasive monitoring device which emits ultra low frequency currents (1.3-14.28 Hz, depending on the programme), low intensity (0.1-0.9 mA), and low voltage (±3 V) and therefore imperceptible to the patient. Each day a different programme was applied. On the first three days, programme 1 (P1) 15 min, programme 2 (P2) 15 min and programme 7 (P7) 30 min were applied. From the fourth to the sixth day, P2 30 min and P7 30 min were applied, finishing the rest of the days with P3 30 min and P7 30 min. At the same time pelvic exercises were performed.
  Interventions: Device: Non-invasive neuromodulation NESA(NNG)
- Group 2: Non Invasive Posterior Tibial Neuromodulation (NTPG) (Active Comparator): Group 2: Non-invasive posterior tibial neuromodulation (NTPG) with same-day exercises and education through common, non-individualised written instructions.
  NTPG was performed by posterior tibial application plus pelvic exercises (same day of treatment) and advice, with the patient supine, using NEUROTRAC MYOPLUS PRO (brand name of the tibial stimulation device) to perform TENS (transcutaneous electric nerve stimulation) for 30 minutes. An electric current with a frequency of 10 Hz and pulse duration of 200μs was applied. The intensity was adjusted according to the patient's tolerance, with thumb flexion perceptible to visual inspection by the therapist. Two 50 x 50 millimeters electrodes were placed along the posterior tibial nerve pathway, one on the sole of the foot and the other near the medial malleolus on one leg.
  Interventions: Device: Non-invasive Neuromodulation Posterior Tibial (NTPG)

INTERVENTIONS:
Device: Non-invasive neuromodulation NESA(NNG) — NESA is a non-invasive monitoring device, which emits low frequency (1.3-14.28 Hz, depending on the programme), low intensity (0.1-0.9 mA), low voltage (±3 V) ultra low currents, and therefore imperceptible to the patient. It is based on neuromodulation of the autonomic nervous system.
  Other Names: NESA neuromodulation; NESA ultra low currents
  Arms: Group1: Non-invasive neuromodulation NESA (NNG group)
Device: Non-invasive Neuromodulation Posterior Tibial (NTPG) — NTPG is an electrotherapy using a device called NEUROTRAC MYOPLUS PRO (brand name) to perform non-invasive TENS-type electrotherapy with biphasic currents.
  Other Names: NEUROTRAC MYOPLUS PRO
  Arms: Group 2: Non Invasive Posterior Tibial Neuromodulation (NTPG)

SUMMARY:
Introduction: Overactive bladder (OAB) is a common condition characterized by urinary urgency, frequency, and, in some cases, urge incontinence. Non-invasive neuromodulation has emerged as an effective therapeutic option by modulating the neural pathways involved in bladder control. This approach offers a promising alternative for patients who do not respond to conventional treatments.

Objectives: To evaluate the effect of non-invasive NESA neuromodulation compared to posterior tibial stimulation in patients with overactive bladder.

compared to posterior tibial stimulation, with same-day exercises and patient education on quality of life, symptoms, discomfort and sleep.

day of the session and patient education on quality of life, symptoms, discomfort and sleep.

Methods: Twenty-four patients (24 women), aged 38-85 years with overactive bladder will be included in this experimental clinical trial study. Each patient will attend ten sessions two days a week. Patient life quality will be measured using SF-36, sleep quality with the Pittsburgh questionnaire, perception of urinari incontinence (UI) symptoms and patient quality of life with the ICIQ-SF questionnaire. All these variables will be measured before, immediately after the ten sessions and at two months after the end of treatment.

Ethic: The study was approved by the ethics committee of the University of Valencia, and all participants will be given an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Minimum criteria for a primary diagnosis of overactive bladder who have or have not received active/alternative treatments for this pathology.
* Patients with previous pharmacological treatments that have not obtained an adequate clinical response.
* Patients whose cognitive abilities are competent to participate in the study and are able to complete the study questionnaires and have given written consent to participate in the study.
* Without further contraindications for electrotherapy treatment such as serious use of pacemakers, pregnancy, internal bleeding, poor skin condition (ulcerations, wounds...) and/or phobia of electricity.

Exclusion Criteria:

* Presence of urinary fistula.
* Infections in the last 12 months.
* Haematuria during the trial period.
* Pregnancy or plans to become pregnant during the study.
* Pathology of the central or peripheral nervous system (multiple sclerosis, Parkinson's disease, etc.).
* Uncontrolled diabetes.
* Currently treated with Botox injections for the bladder or within the last year.
* Current treatment with interstim or currently implanted interstim device.
* Bladder outlet obstruction.
* Urinary retention.
* Treatment with more than two antidepressants and/or multiple benzodiazepines, as well as antiepileptics.
* Contraindications for electrotherapy treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 questionnaire | Before treatment, immediately after the treatment is finished and at two months later (follow-up)
  The SF-36 is a 36-question survey that assesses health-related quality of life, measuring eight key domains: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems, and mental health. It's a widely used tool in clinical practice and research for evaluating health status and assessing the impact of interventions.

SECONDARY OUTCOMES:
Pittsburgh questionnaire | Sleep quality was assessed before, immediately after and at two months
  Sleep quality using the Pittsburgh questionnaire, consisting of 19 items that analyse 7 different components of sleep (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction). Each item is scored from 0 to 3. The total score of the scale ranges from 0 to 21 points where the lower end represents good sleep quality, and the upper end represents poor sleep quality
ICIQ-UI Short Form | ICIQ-SF was assessed before treatment, immediately after the treatment is finished and at two months later (follow-up)
  Perception of frequency, severity of urinary incontinence (UI) and patient quality of life were assessed using the International Consultation on Incontinence Questionnaire (ICIQ-SF) validated questionnaire, where the individual's daily experience of urination and incontinence is answered with three scored items and one unmarked self-diagnostic item.
Bladder Control Self-Assessment Questionnaire (B-SAQ) | Before treatment, immediately after the treatment is finished and at two months later (follow-up)
  Bladder symptoms and discomfort were assessed using the Bladder Control Self-Assessment Questionnaire (B-SAQ), a validated questionnaire consisting of 8 questions grouped into two scales, each with a scale of 0 to 3 points, giving a maximum score of 24 points (12 in each group).
Personal satisfaction of patients | In the follow-up (two month later)
  After two months they were asked about their satisfaction with the treatment received (numerical scale from 0 not satisfied -10 very satisfied), whether they continued to do the exercises and whether they had any side effects after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Blasco-Sonora, Physical Therapy, Principal Investigator — University of Valencia; Laura FUENTES-APARICIO, PhD. Physical Therapy, Study Director — University of Valencia; Raquel Medina-Ramírez, PhD. Physical Therapy, Study Director — University of Las Palmas
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Not to be shared

REFERENCES:
- [Background] Teruel-Hernandez E, Lopez-Pina JA, Souto-Camba S, Baez-Suarez A, Medina-Ramirez R, Gomez-Conesa A. Improving Sleep Quality, Daytime Sleepiness, and Cognitive Function in Patients with Dementia by Therapeutic Exercise and NESA Neuromodulation: A Multicenter Clinical Trial. Int J Environ Res Public Health. 2023 Nov 6;20(21):7027. doi: 10.3390/ijerph20217027. PMID 37947583
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Lo CW, Wu MY, Yang SS, Jaw FS, Chang SJ. Comparing the Efficacy of OnabotulinumtoxinA, Sacral Neuromodulation, and Peripheral Tibial Nerve Stimulation as Third Line Treatment for the Management of Overactive Bladder Symptoms in Adults: Systematic Review and Network Meta-Analysis. Toxins (Basel). 2020 Feb 18;12(2):128. doi: 10.3390/toxins12020128. PMID 32085542
- [Background] Przydacz M, Golabek T, Dudek P, Lipinski M, Chlosta P. Prevalence and bother of lower urinary tract symptoms and overactive bladder in Poland, an Eastern European Study. Sci Rep. 2020 Nov 13;10(1):19819. doi: 10.1038/s41598-020-76846-0. PMID 33188254

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT07019597/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT07019597/ICF_001.pdf